CLINICAL TRIAL: NCT00920777
Title: A RCT Study on the Effect of Short and Long Cognitive Behaviour Therapy (CBT) in CFS/ME Patients
Brief Title: Survey and Cognitive Behavior Therapy for Chronic Fatigue Syndrome/Myalgic Encephalomyelitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 21592; 21592 (Other: NSD); 4.2008.2586 (Other: REK)
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Chronic Fatigue Syndrome; Myalgic Encephalomyelitis; Fatigue; Pain
Keywords: CBT; Fukuda criteria; Mental functioning; Physical functioning
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Fatigue; Pain | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 8 weeks CBT (Experimental)
  Interventions: Behavioral: CBT
- Control group (Active Comparator)
  Interventions: Behavioral: Control group
- 16 weeks CBT (Experimental)
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: CBT — Individual Cognitive Behavior Therapy during 16 weeks
  Other Names: Grades excercise therapy
  Arms: 16 weeks CBT
Behavioral: CBT — Individual Cognitive Behavior Therapy during 8 weeks
  Arms: 8 weeks CBT
Behavioral: Control group — Waiting 16 weeks and receiving 8 weeks individual CBT after waiting period.
  Arms: Control group

SUMMARY:
The purpose of this study is to analyze income variables in Chronic Fatigue Syndrome/Myalgic Encephalomyelitis, and to analyze the effect of short vs. long Cognitive Behaviour Therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to St.Olav Hospital, Trondheim
* fulfil the FUKUDA criteria for CFS/ME.

Exclusion Criteria:

* Pregnant patients

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 234 (Actual)
Dates: Start 2009-05; Primary Completion 2014-07 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Mental and physical function | 1 year
  Mental and physical function, measured by "SF 36". Success criteria are measured by >10 point improvement of mental and/ or physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Egil Fors, prof MD, Principal Investigator — St. Olavs Hospital
Locations (1):
- St.Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Rasouli O, Gotaas ME, Stensdotter AK, Skovlund E, Landro NI, Dastol P, Fors EA. Neuropsychological dysfunction in chronic fatigue syndrome and the relation between objective and subjective findings. Neuropsychology. 2019 Jul;33(5):658-669. doi: 10.1037/neu0000550. Epub 2019 Jun 6. PMID 31169386
- [Derived] Gotaas ME, Stiles TC, Bjorngaard JH, Borchgrevink PC, Fors EA. Cognitive Behavioral Therapy Improves Physical Function and Fatigue in Mild and Moderate Chronic Fatigue Syndrome: A Consecutive Randomized Controlled Trial of Standard and Short Interventions. Front Psychiatry. 2021 Apr 12;12:580924. doi: 10.3389/fpsyt.2021.580924. eCollection 2021. PMID 33912079